CLINICAL TRIAL: NCT00964587
Title: Randomized Trial of CVD Education and Problem-Solving Training in Urban Diabetics
Brief Title: Cardiovascular Disease Education and Problem-Solving Training in People With Type 2 Diabetes
Acronym: DECIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Felicia Hill-Briggs, Assoc. Professor of Medicine, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HL089751-01A1 (NIH); R01HL089751-01A1 (NIH)
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes
Keywords: diabetes self management education; problem-solving training; health behavior change; health literacy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Usual Care (Active Comparator): Packet of standard print patient education materials on CVD and diabetes from the American Heart Association (AHA) and the American Diabetes Association (ADA).
  Interventions: Behavioral: Usual Care
- Self Study (Experimental): One 90-minute educational session. Print materials and DVDs for self-study
  Interventions: Behavioral: Education + Problem-Solving Training Self-Study
- Group Problem-Solving Training (Experimental): One 90-minute education session. Group problem-solving training (eight, 90-minute sessions)
  Interventions: Behavioral: Education + Group Problem-Solving Training
- Individual Problem-Solving Training (Experimental): One 90-minute education session. Individual problem-solving training (eight, 60-minute sessions)
  Interventions: Behavioral: Education + Individual Problem-Solving Training

INTERVENTIONS:
Behavioral: Education + Problem-Solving Training Self-Study — * Education + Problem-Solving Training Self-Study
  * One session of Literacy-Adapted Diabetes and CVD Risk Education
  * Instructions and a schedule for use of the Literacy-Adapted Problem-Solving Workbook for self-study will be given to each participant.
  Other Names: Self-Management Training Self-Study; Project DECIDE Self-Study
  Arms: Self Study
Behavioral: Education + Group Problem-Solving Training — * Education + Group Problem-Solving Training
  * One session of the Literacy-Adapted Diabetes and CVD Risk Education
  * Group problem-solving training eight, 90-minute sessions
  Other Names: Group Self-Management Training; Project DECIDE Group Training
  Arms: Group Problem-Solving Training
Behavioral: Education + Individual Problem-Solving Training — * Education + Individual Problem-Solving Training
  * One session of the Literacy-Adapted Diabetes and CVD Risk Education
  * Individual problem-solving training (eight, 60-minute sessions)
  Other Names: Individual Self-Management Training; Project DECIDE Individual Training
  Arms: Individual Problem-Solving Training
Behavioral: Usual Care — * Packet of print patient education materials about CVD and diabetes from the American Heart Association (AHA) and the American Diabetes Association (ADA)given at baseline following randomization to Arm 1
  * Scripted set of instructions will be given along with a verbal description of the materials and the content provided.
  Other Names: Standard Print Education Materials; Project DECIDE Usual Care
  Arms: Usual Care

SUMMARY:
The purpose of this study is to determine if patient education and problem-solving training, delivered in self-study, group, and individual intervention modalities, will produce substantial improvements in CVD risk profile via improved self management in urban African Americans with type 2 diabetes and a high CVD risk profile.

DETAILED DESCRIPTION:
African Americans with type 2 diabetes suffer excess disease burden, but cardiovascular disease (CVD) risk factors such as hyperglycemia, hypertension, and dyslipidemia are modifiable with medical management and lifestyle modification. Patient diabetes education and counseling for behavior change are recommended standards of practice to facilitate effective self-management of these risk factors. However, for patients with low literacy or health literacy, accessibility and impact of educational and behavioral interventions are limited. Pilot research suggests that: a) literacy demand and behavioral activation characteristics of patient education modules can be adapted to facilitate learning in urban patients with low literacy, and b) combining literacy-adapted education with problem-solving training facilitates understanding and use of health information for performing self-management in the context of daily life (functional health literacy). Optimal modalities for delivery of a combined patient diabetes education and problem-solving training, and cost-effectiveness of this intervention model, however, are not known. The proposed study will address these needs by testing effectiveness and cost-effectiveness of literacy-adapted diabetes and CVD education and problem-solving training interventions in urban African Americans with type 2 diabetes and high CVD risk profile (suboptimal blood sugar, blood pressure, and/or lipids). The specific aims of the study are: a) to complete development of a package of literacy-adapted diabetes and CVD patient education materials by developing two video/DVDs addressing self-management recommendations appropriate to the needs, resources, and environment of the population; b) to randomize urban African-American adults with type 2 diabetes and a high CVD risk profile into one of four study arms: Usual Care (Arm 1), Literacy-Adapted Education and Problem-Solving Training Self-Study (Arm 2), Literacy-Adapted Education and Group Problem-Solving Training (Arm 3), and Literacy-Adapted Education and Individual Problem-Solving Training (Arm 4); c) to conduct baseline, 3-month post-intervention, and 6-month post-intervention assessment visits to analyze and compare effectiveness of the literacy-adapted education and problem-solving interventions, as compared to Usual Care, in improving the skills of knowledge, problem-solving and health literacy, behaviors of patient activation and diabetes self-management, and clinical outcomes of A1C, blood pressure and lipids; and d) to perform a cost-effectiveness analysis of each intervention arm as compared to Usual Care. If proven effective, this research will yield low literacy diabetes and CVD patient education and self-management intervention tools for dissemination to high-risk urban minority populations. Moreover, the cost-effectiveness analysis will provide evidence to support decision-making regarding implementation of the models to achieve cardiovascular disease patient self-management goals in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 years or older

  * Type 2 diabetes determined by physician diagnosis or self-report of type 2 diabetes confirmed by medical documentation or medication review
  * Black/African American by self-report
  * currently receiving care and able to provide contact information for a treating physician
  * residing in Baltimore, Maryland.

Exclusion Criteria:

* Mentally incompetent to give informed consent
* Severe cognitive impairment on the Telephone Interview for Cognitive Status
* Unable to complete assessment (interview, tests, venipuncture)
* Comorbid conditions likely to lead to death in the next 3-5 years (e.g. cancer, AIDS, end-stage renal disease, active tuberculosis, Alzheimer's disease)
* Planning to relocate from Baltimore region during the time period of the study or other reasons rendering person unable to attend visits to participate in intervention and follow-up assessments

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2010-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
HbA1C | Screening, 3 months post intervention, 6 months post-intervention

SECONDARY OUTCOMES:
Blood pressure | Screening, 3 months post-intervention, 6 months post-intervention
Lipid Panel | Screening, 3 months post-intervention, 6 months post-intervention
Body Mass Index | Screening, 3 months post-intervention, 6 months post-intervention
Health Problem Solving Scale | Screening, 1 week post-intervention, 3 months post-intervention, 6 months post-intervention
Diabetes and CVD Knowledge Test | Screening, 3 months post-intervention, 6 months post-intervention
Patient Activation Measure | Baseline, 3 months post-intervention, 6 months post-intervention
Summary of Diabetes Self-Care Activities Scale | Baseline, 3 months post-intervention, 6 months post-intervention
Barriers to Self-Management | Baseline, 1 week post-intervention, 3 months post-intervention, 6 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Hill-Briggs, PhD, ABPP, Principal Investigator — Johns Hopkins School of Medicine
Locations (3):
- United States (3):
  - Johns Hopkins School of Medicine/General Clinical Research Center, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center/General Clinical Research Center, Baltimore, Maryland
  - Johns Hopkins School of Medicine/General Internal Medicine, Baltimore, Maryland

REFERENCES:
- [Background] Hill-Briggs F, Gemmell L. Problem solving in diabetes self-management and control: a systematic review of the literature. Diabetes Educ. 2007 Nov-Dec;33(6):1032-50; discussion 1051-2. doi: 10.1177/0145721707308412. PMID 18057272
- [Background] Hill-Briggs F, Smith AS. Evaluation of diabetes and cardiovascular disease print patient education materials for use with low-health literate populations. Diabetes Care. 2008 Apr;31(4):667-71. doi: 10.2337/dc07-1365. Epub 2008 Jan 17. PMID 18202245
- [Background] Hill-Briggs F, Gemmell L, Kulkarni B, Klick B, Brancati FL. Associations of patient health-related problem solving with disease control, emergency department visits, and hospitalizations in HIV and diabetes clinic samples. J Gen Intern Med. 2007 May;22(5):649-54. doi: 10.1007/s11606-006-0091-2. PMID 17443373
- [Background] Hill-Briggs F. Problem solving in diabetes self-management: a model of chronic illness self-management behavior. Ann Behav Med. 2003 Summer;25(3):182-93. doi: 10.1207/S15324796ABM2503_04. PMID 12763713
- [Background] Hill-Briggs F, Renosky R, Lazo M, Bone L, Hill M, Levine D, Brancati FL, Peyrot M. Development and pilot evaluation of literacy-adapted diabetes and CVD education in urban, diabetic African Americans. J Gen Intern Med. 2008 Sep;23(9):1491-4. doi: 10.1007/s11606-008-0679-9. Epub 2008 Jun 3. PMID 18521688
- [Background] Majid HM, Schumann KP, Doswell A, Sutherland J, Hill Golden S, Stewart KJ, Hill-Briggs F. Development and evaluation of the DECIDE to move! Physical activity educational video. Diabetes Educ. 2012 Nov-Dec;38(6):855-9. doi: 10.1177/0145721712462748. Epub 2012 Oct 4. PMID 23042504
- [Background] Hill-Briggs F, Schumann KP, Dike O. Five-step methodology for evaluation and adaptation of print patient health information to meet the < 5th grade readability criterion. Med Care. 2012 Apr;50(4):294-301. doi: 10.1097/MLR.0b013e318249d6c8. PMID 22354210
- [Background] Fitzpatrick SL, Schumann KP, Hill-Briggs F. Problem solving interventions for diabetes self-management and control: a systematic review of the literature. Diabetes Res Clin Pract. 2013 May;100(2):145-61. doi: 10.1016/j.diabres.2012.12.016. Epub 2013 Jan 9. PMID 23312614
- [Derived] Fitzpatrick SL, Golden SH, Stewart K, Sutherland J, DeGross S, Brown T, Wang NY, Allen J, Cooper LA, Hill-Briggs F. Effect of DECIDE (Decision-making Education for Choices In Diabetes Everyday) Program Delivery Modalities on Clinical and Behavioral Outcomes in Urban African Americans With Type 2 Diabetes: A Randomized Trial. Diabetes Care. 2016 Dec;39(12):2149-2157. doi: 10.2337/dc16-0941. PMID 27879359